CLINICAL TRIAL: NCT06143046
Title: A Phase 2, Randomized, Observer-Blind, Placebo-Controlled, Dose-Escalation Study to Evaluate the Reactogenicity, Safety, and Immunogenicity of mRNA-1345, an mRNA Vaccine Targeting Respiratory Syncytial Virus, in Pregnant Women, and Safety and Immunogenicity in Infants Born to Vaccinated Mothers
Brief Title: A Study of mRNA-1345 Vaccine Targeting Respiratory Syncytial Virus in Pregnant Women and in Infants Born to Vaccinated Mothers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: mRNA-1345-P201; 2023-505359-37-00 (Other: EU CT number)
Record Dates: First submitted 2023-11-14; First posted 2023-11-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Respiratory Syncytial Virus
Keywords: mRNA-1345; RSV vaccine; Viral Diseases; Messenger RNA; Moderna
MeSH Terms: conditions — Virus Diseases | interventions — mRNA-1345 respiratory syncytial virus vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- mRNA-1345 Dose A (Experimental): Participants will be vaccinated in the period from 28 weeks to 36 weeks of gestation with a single intramuscular (IM) injection of mRNA-1345 Dose A.
  Interventions: Biological: mRNA-1345
- mRNA-1345 Dose B (Experimental): Participants will be vaccinated in the period from 28 weeks to 36 weeks of gestation with a single IM injection of mRNA-1345 Dose B.
  Interventions: Biological: mRNA-1345
- mRNA-1345 Dose C (Experimental): Participants will be vaccinated in the period from 28 weeks to 36 weeks of gestation with a single IM injection of mRNA-1345 Dose C.
  Interventions: Biological: mRNA-1345
- Placebo (Placebo Comparator): Participants will receive single IM injection of mRNA-1345 vaccine matching placebo in the period from 28 weeks to 36 weeks of gestation.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: mRNA-1345 — Sterile liquid for injection
  Arms: mRNA-1345 Dose A; mRNA-1345 Dose B; mRNA-1345 Dose C
Biological: Placebo — 0.9% sodium chloride (normal saline) injection
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate the reactogenicity, safety, and immunogenicity of an investigational respiratory syncytial virus (RSV) vaccine, mRNA-1345, in pregnant women, and safety and immunogenicity in infants born to vaccinated mothers.

ELIGIBILITY:
Key Inclusion Criteria:

Maternal Participants

* Are adults ≥18 years to <40 years of age inclusive, at the time of signing the informed consent.
* Will be 28 to 36 weeks pregnant at the time of vaccination (confirmed by an obstetric ultrasound report).
* Intend to deliver at a maternity unit where study procedures can be performed.
* Are willing and able to attend all study visits, to undergo all study procedures/or have their infant undergo all study procedures, and to comply with study requirements, including a means of communication (for example, phone, text message or email) with study site staff.
* Have engaged with local antenatal care and will continue to do so through the remainder of their pregnancy.
* Have had an antenatal obstetric ultrasound at ≥18 weeks of pregnancy or be willing to have an antenatal obstetric ultrasound at Screening if not already conducted.

Specific inclusion criteria for Japanese pregnant women:

* Japanese participants are defined as individuals born in Japan, with both parents and 4 grandparents who were born in Japan.

Infant Participants

* Have consent from infant participant's parent(s)/legally authorized representative (LAR) if required by local regulations.

Key Exclusion Criteria:

Maternal Participants

* Acutely ill or febrile (temperature ≥38.0 degrees Celsius [℃]/100.4 degrees Fahrenheit [°F]) within 72 hours prior to or at the Screening Visit or Day 1.
* Reported history of anaphylaxis or severe hypersensitivity reaction after receipt of any mRNA vaccine or therapeutic or any components of an mRNA-1345 vaccine.
* Any medical, psychiatric, or occupational condition, including reported history of drug or alcohol abuse, that, in the opinion of the Investigator, might pose additional risk due to participation in the study or could interfere with the interpretation of study results.
* Have conditions in the current pregnancy or in previous pregnancies that may affect participant safety, assessment of safety endpoints, assessment of immune response, or adherence to study procedures.
* Received or plans to receive any mRNA vaccine or COVID-19 vaccine within 4 weeks before or after Day 1 and/or any other nonstudy vaccine within 2 weeks before or after Day 1.
* Previous vaccination with any licensed or investigational RSV vaccine or planned receipt during study participation.
* Intend for their infant to receive RSV monoclonal antibodies after delivery.

Infant Participants

* Is a child who has been placed under the control or protection of an agency, organization, institution, or entity by the courts, the government, or a government body acting in accordance with powers conferred on them by laws and regulation (for example, foster care). This does not include a child who is adopted or has an appointed LAR.

Other inclusion and exclusion criteria may apply.

Ages: 0 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 360 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2026-05-27 (Estimated); Study Completion 2026-05-27 (Estimated)

PRIMARY OUTCOMES:
Number of Maternal Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 7 (7 days post vaccination)
Number of Maternal Participants with Unsolicited Adverse Events (AEs) | Up to Day 28 (28 days post vaccination)
Number of Maternal Participants with Medically-Attended AEs (MAAEs) | Day 1 to Month 6 (6 months postdelivery)
Number of Maternal Participants with Adverse Events of Special Interest (AESIs) | Day 1 to Month 12 (12 months postdelivery)
Number of Maternal Participants with Serious Adverse Events (SAEs) | Day 1 to Month 12 (12 months postdelivery)
Number of Maternal Participants with AEs Leading to Discontinuation | Day 1 to Month 12 (12 months postdelivery)
Number of Maternal Participants With Pregnancy Outcomes | Day 1 to Month 12 (12 months postdelivery)
  Pregnancy outcomes will include stillbirth, live birth, vaginal delivery, and cesarean section delivery.
Number of Infant Participants with MAAEs | Day 1 (birth) to Month 12
Number of Infant Participants with AESIs | Day 1 (birth) to Month 12
Number of Infant Participants with SAEs | Day 1 (birth) to Month 12
Number of Infant Participants With Birth Outcomes | Day 1 (birth) to Month 12
  Birth outcomes will include gestational age and anthropometric measurements.

SECONDARY OUTCOMES:
Geometric Mean Titer (GMT) of Serum RSV-A and RSV-B Neutralizing Antibodies in Maternal Participants | Day 1, Day 29, delivery, and Month 6 (6 months postdelivery)
Geometric Mean Concentration (GMC) of Serum RSV-F Binding Antibodies in Maternal Participants | Day 1, Day 29, delivery, and Month 6 (6 months postdelivery)
Geometric Mean Fold-Rise (GMFR) of Postbaseline/Baseline Neutralizing Antibody Titers and Binding Antibody Concentrations in Maternal Participants | Day 29, delivery, and Month 6 (6 months postdelivery)
Percentage of Maternal Participants With ≥4-fold Increase From Baseline in Neutralizing Antibody Titers and Binding Antibody Concentrations | Baseline up to Month 6 (6 months postdelivery)
GMT of Serum RSV-A and RSV-B Neutralizing Antibodies in Infant Participants | Day 1 (birth), and Months 2, 6, and 12
GMC of Serum RSV-F Binding Antibodies in Infant Participants | Day 1 (birth), and Months 2, 6, and 12

CONTACTS AND LOCATIONS:
Locations (56):
- United States (22):
  - SEC Clinical Research LLC - Dothan 2 - ClinEdge - PPDS, Dothan, Alabama
  - Abby's Research Institute, Phoenix, Arizona
  - Watching Over Mothers & Babies, Tucson, Arizona
  - Applied Research Center of Arkansas - ClinEdge - PPDS, Little Rock, Arkansas
  - Matrix Clinical Research - Gardena, Gardena, California
  - Matrix Clinical Research - Huntington Park, Huntington Park, California
  - Matrix Clinical Research, Inc - Corporate Office, Los Angeles, California
  - Clinical Research Prime - ClinEdge - PPDS, Idaho Falls, Idaho
  - Bingham Memorial Hospital, Pocatello, Idaho
  - Clinical Research Prime - ClinEdge - Rexburg - PPDS, Rexburg, Idaho
  - Velocity Clinical Research - Covington - PPDS, Covington, Louisiana
  - Saginaw Valley Medical Research Group LLC, Saginaw, Michigan
  - Boeson Research GTF - Great Falls - ERN - PPDS, Great Falls, Montana
  - Boeson Research KAL - Kalispell - ERN - PPDS, Kalispell, Montana
  - Boeson Research MSO - Missoula - ERN - PPDS, Missoula, Montana
  - Velocity Clinical Research (Grand Island - Nebraska) - PPDS, Grand Island, Nebraska
  - Velocity Clinical Research (Hastings - Nebraska) - PPDS, Hastings, Nebraska
  - Velocity Clinical Research (Norfolk - Nebraska) - PPDS, Norfolk, Nebraska
  - DM Clinical Research - Bellaire - ERN - PPDS, Houston, Texas
  - Maximos OB/GYN, League City, Texas
  - SMS Clinical Research, Mesquite, Texas
  - Maternal Fetal Diagnostics Center, Salt Lake City, Utah
- Canada (4):
  - Dalhousie University - 5820 University Ave, Halifax, Nova Scotia
  - Ottawa Hospital, Ottawa, Ontario
  - Sainte Justine Hospital, Montreal, Quebec
  - Centre Hospitalier de l'Université Laval, Québec
- Chile (3):
  - Clínica Universidad de los Andes, Las Condes, Región-MetropolitanadeSantiago
  - Centro Internacional de Estudios Clínicos, Recoleta, Región-MetropolitanadeSantiago
  - Red Hospital Clinico de la Universidad de Chile, Santiago
- Denmark (3):
  - Hvidovre Hospital, Hvidovre, Capital
  - Aarhus Universitetshospital, Aarhus, Central Jutland
  - Regionshospitalet Gødstrup, Herning, Central Jutland
- Japan (4):
  - Shonan Kamakura General Hospital, Kamakura-Shi, Kanagawa
  - Saiseikai Yokohamashi Nanbu Hospital, Yokohama, Kanagawa
  - Saitama City Hospital, Saitama-Shi, Saitama
  - Center Hospital of the National Center for Global Health and Medicine, Shinjuku-Ku, Tokyo
- Panama (5):
  - Centro De Vacunacion Internacional, S.A. (Cevaxin) - David, David, Chiriquí Province
  - Centro De Vacunacion Internacional, S.A. (Cevaxin) Sede La Chorrera, Panama City
  - Centro De Vacunacion Internacional, S.A. (Cevaxin), Panama City
  - CEVAXIN 24 de diciembre, Panama City
  - Instituto de Investigaciones Científicas Y Servicios de Alta Tecnología Asociación de Interés Panama, Pueblo Nuevo
- South Africa (8):
  - Josha Research, Bloemfontein, Free State
  - Drs. YAK Vahed & Partners, Welkom, Free State
  - Ubuntu Clinical Research, Krugersdorp, Gauteng
  - Bothe ke Bontle Health Services-316 Kuit st, Pretoria, Gauteng
  - Setshaba Research Centre, Soshanguve, Gauteng
  - WITS Clinical Research Site - PPDS, Soweto, Gauteng
  - Merclinico Middelburg, Middelburg, Mpumalanga
  - FAM-CRU, Cape Town, Western Cape
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Southampton General Hospital, Southampton, Hampshire
  - The Royal London Hospital, London, London, City of
  - The Royal Free Hospital, London, Middlesex
  - Cardiff & Vale University Health Board-PPDS, Cardiff, South Glamorgan
  - St George's Hospital, London, Surrey
  - Glasgow Clinical Research Facility - PPDS, Glasgow